CLINICAL TRIAL: NCT05035641
Title: A Pilot Phase II Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled, Dose-Ranging, Safety and Efficacy Study of Oral AND017 to Treat Anemia in Nondialysis-Dependent Chronic Kidney Disease (NDD-CKD) Patients
Brief Title: A Study of AND017 to Treat Anemia in Non-dialysis-Dependent Chronic Kidney Disease (NDD-CKD) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kind Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AND017-MN-201
Record Dates: First submitted 2021-04-21; First posted 2021-09-05 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Renal Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AND017 Dose A (Experimental): AND017 will be administrated orally at dose A
  Interventions: Drug: AND017
- AND017 Dose B (Experimental): AND017 will be administrated orally at dose B
  Interventions: Drug: AND017
- AND017 Dose C (Experimental): AND017 will be administrated orally at dose C
  Interventions: Drug: AND017
- Placebo (Placebo Comparator): Placebo will be administrated orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AND017 — Orally, 3 times per week in Period 1 and randomize to TIW or QW group at the same dose in Period 2
  Arms: AND017 Dose A; AND017 Dose B; AND017 Dose C
Drug: Placebo — Orally, 3 times per week
  Arms: Placebo

SUMMARY:
This is a pilot phase II study to evaluate the safety and efficacy of AND017 in NDD-CKD patients

DETAILED DESCRIPTION:
This is a pilot phase 2, multicenter, randomized, parallel-group, double-blind, placebo-controlled, dose-ranging, safety and efficacy study of oral AND017 to treat anemia in non-dialysis-dependent chronic kidney disease patients.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of chronic kidney disease, not receiving dialysis, with an eGFR <60 mL/min/1.73 m2.
2. Baseline Hb level ≥ 7.5 g/dL and <10.0 g/dL.
3. TSAT ≥ 20% or ferritin ≥ 100 ng/mL at screening test
4. Serum folate and vitamin B12 ≥ lower limit of normal at screening test
5. AST and ALT ≤ 3×ULN.
6. Total bilirubin ≤ 1.5×ULN.

Key Exclusion Criteria:

1. Concurrent retinal neovascular lesions requiring treatment including proliferative diabetic retinopathy, exudative age-related macular degeneration, retinal vein occlusion, macular edema, etc.
2. Anemia that is possibly mainly caused by concurrent autoimmune disease with inflammatory symptoms
3. History of gastric/intestinal resection considered to affect the absorption of drugs in the gastrointestinal tract (excluding resection of gastric or colon polyps) or concurrent symptomatic gastroparesis despite being on treatment.
4. Clinically significant bleeding (eg, requiring transfusion or drop in Hb of ≥ 2g/dL) within 4 weeks of first dose; no bleeding diathesis or risk of bleeding that has not been medically or surgically corrected at least 4 weeks prior to first dose of study drug.
5. Uncontrolled hypertension defined as patients with hypertension having more than one of three diastolic blood pressure values >95 mmHg and each test at least 5 min apart during the screening assessment.
6. Concurrent congestive heart failure (New York Heart Association [NYHA] Class III or higher).
7. History of stroke, transient ischemic attack, myocardial infarction, thromboembolic event, pulmonary embolism, or lung infarction within 24 weeks before the screening assessment.
8. Concurrent anemia due to another cause other than renal anemia
9. Known hemosiderosis, hemochromatosis or hyper-coagulable condition
10. Any treatment with a hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI) within 5 weeks before randomization.
11. Having received treatment with erythropoiesis stimulating agents, androgenic anabolic steroids, testosterone enanthate, or mepitiostane within 5 weeks before the first dose.
12. Total bilirubin >1.5xULN, or AST>3xULN, or ALT>3xULN, or ALP>3xULN, or previous or concurrent serious liver disease (acute or active chronic hepatitis, cirrhosis, etc.) thought to be caused by ESAs.
13. Patients with a history of significant liver disease or active liver disease. Investigators should discuss this with the Medical Monitor for cases where there is doubt about whether to exclude or not.

13. Patients that have major surgery planned during the study period. 14. Having undergone blood transfusion and/or a surgical procedure within 8 weeks before the screening assessment.

15. Having undergone a kidney transplantation. 16. History of a seizure disorder or any occurrence of seizures in the past

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Safety Evaluations | Up to 17 weeks
  Incidence of adverse events
Rate of rise in hemoglobin for each of 3 dose levels as compared with placebo from baseline to 5 weeks after TIW oral dosing | Up to 5 weeks after dosing
  Calculate the slope of a linear regression for each patient using all hemoglobin data collected during the Fixed-Dose Period

SECONDARY OUTCOMES:
Hb response to treatment during Period 1 | Up to 5 weeks after dosing
  Cumulative percentage of patients with Hb ≥10.0 g/dL
Percentage of responder patients | Up to 13 weeks after dosing
  Responder is defined as a hemoglobin ≥10.0 g/dL and an increase in hemoglobin by ≥1.0 g/dL
Percentage of visits at which patients maintain hemoglobin between 10.0-11.0 g/dL after achieving hemoglobin ≥10.0 g/dL | Up to 13 weeks after dosing
  Percentage of visits at which patients maintain hemoglobin between 10.0-11.0 g/dL after achieving hemoglobin ≥10.0 g/dL
Change from baseline in Hb | Up to 13 weeks after dosing
  Change from baseline in Hb
Change in hemoglobin levels from baseline to the mean of weeks 10-13 | Baseline and at Week 10, 11, 12, 13, and 14
  Change in hemoglobin levels from baseline to the mean of weeks 10-13
Percentage of patients who maintain hemoglobin between 10.0-11.0g/dL at each visit | Up to 13 weeks after dosing
  Percentage of patients who maintain hemoglobin between 10.0-11.0g/dL at each visit
Mean Hb levels at weeks 6-14 including the average of weeks 10-13 | Up to 13 weeks after dosing
  Mean Hb levels at weeks 6-14 including the average of weeks 10-13
Cumulative incidence of lack of response over the entire treatment period | Up to13 weeks after dosing
  Hb level < 10.0 g/dL and an increase in hemoglobin from baseline of < 1 g/dL
To assess changes in the levels of PD indicator - EPO | Baseline and at Week 2, 4, 6, 8, 10, 12, 14, and 28 days after the last dose
  To assess changes in the levels of EPO
To assess changes in the levels of PD indicator - hepcidin | Baseline and at Week 2, 4, 6, 8, 10, 12, 14, and 28 days after the last dose
  To assess changes in the levels of hepcidin
To assess iron utilization parameter during treatment - transferrin level | Baseline and at Week 3, 6, 9, 12, 14, and 28 days after the last dose
  To assess transferrin level during treatment
To assess iron utilization parameter during treatment - total iron-binding capacity (TIBC) | Baseline and at Week 3, 6, 9, 12, 14, and 28 days after the last dose
  To assess TIBC level during treatment
To assess iron utilization parameter during treatment - transferrin saturation (TSAT) | Baseline and at Week 3, 6, 9, 12, 14, and 28 days after the last dose
  To assess TSAT level during treatment
To assess iron utilization parameters during treatment - ferritin | Baseline and at Week 3, 6, 9, 12, 14, and 28 days after the last dose
  To assess ferritin level during treatment
To assess iron utilization parameters during treatment - serum iron | Baseline and at Week 3, 6, 9, 12, 14, and 28 days after the last dose
  To assess serum iron level during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yusha Zhu, MD PhD, Study Director — Kind Pharmaceuticals LLC
Locations (8):
- United States (7):
  - Amicis Research Center, Northridge, California
  - Clinical Site Partners, Winter Park, Florida
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Elite Research Center, Flint, Michigan
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Clinical Advancement Center, PLLC, San Antonio, Texas
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No